CLINICAL TRIAL: NCT06228469
Title: Cytolytic Vaginosis Multicentre Registry
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00122929
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Cytolytic Vaginosis
Keywords: Vaginitis; Lactobacillus; Wet mount; Vaginal microbiome; Fragmented epithelial cells; Vaginal discharge
MeSH Terms: conditions — Vaginitis; Vaginal Discharge

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women diagnosed with cytolytic vaginosis: Women presenting to an outpatient clinic with vaginitis symptoms and diagnosed with cytolytic vaginosis.

SUMMARY:
The goal of this registry is to learn more about cytolytic vaginosis, a little known and controversial condition. The main questions the registry aims to answer are:

* What are risk factors of cytolytic vaginosis?
* Are there defining symptoms of cytolytic vaginosis?
* What features on wet mount should be used to diagnosis cytolytic vaginosis?
* Are baking soda vaginal irrigations an effective treatment for cytolytic vaginosis?
* Do characteristics of cytolytic vaginosis vary between sites/countries?

DETAILED DESCRIPTION:
Cytolytic vaginosis is a largely unknown, debated, and equivocal vaginal condition. It is unclear whether cytolytic vaginosis is a variant of normal vaginal microbiome or should be considered a vaginal dysbiosis condition, similar to bacterial vaginosis. This multicentre registry will enroll women that have signs/symptoms consistent with cytolytic vaginosis to better characterize it.

Women at participating sites diagnosed with cytolytic vaginosis and that provide consent will be consecutively enrolled in the registry. The registry will capture data on risk factors, symptoms, test results (eg, wet mount) and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Vaginitis symptoms
* Predominately lactobacilli or/and elongated lactobacilli on wet mount
* Cytolysis on wet mount

Exclusion Criteria:

* Unable to consent or decline consent
* Pregnant
* Positive for yeast (culture or PCR)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women attending an outpatient clinic with vaginitis symptoms
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Characterize cytolytic vaginosis | 1 year
  Describe the risk factors, symptoms, signs and treatment outcomes of cytoytic vaginosis

CONTACTS AND LOCATIONS:
Locations (3):
- Universidade Federal Fluminense-UFF, Niterói, Rio de Janeiro, Brazil
- Outpatient clinics, Multiple Locations, Alberta, Canada
- Centro Hospitalar de São João, Porto, Portugal